CLINICAL TRIAL: NCT02519465
Title: Evaluation of Lung Deposition of Aerosol Via HFNC in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, Luciana Alcoforado Mendes da Silva, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Luciana doutorado 02
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: nasal cannula; Inhalation Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HEATED FLOW (Active Comparator): The volunteers were randomly allocated into three groups - group 1 - 10l/min cold or heated, group 2 - 30l/min cold or heated, group 3 - 50 l /min - cold or heatedPhase 1 - 10l/min or 30l/min or 50l/min of the oxygen heated .
  Interventions: Other: 10l/min; Other: 30l/min; Other: 50l/min
- COLD FLOW (Active Comparator): The volunteers were randomly allocated into three groups - group 1 - 10l/min cold or heated, group 2 - 30l/min cold or heated, group 3 - 50 l /min - cold or heatedPhase 1 - 10l/min or 30l/min or 50l/min of the oxygen cold
  Interventions: Other: 10l/min; Other: 30l/min; Other: 50l/min

INTERVENTIONS:
Other: 10l/min — For inhalation was used diethilene penta-acetic triamine technetium (99mTc-DTPA) with radioactivity of 1 millicuries (Noble et al., 2007) and 0.9% saline solution with a total volume of 1 ml using vibrating mesh inhaler (Aerogen Ltd, Galway , Ireland) with the respiratory care system for the high flow ( Fisher & Paykel healthcare, New Zealand) and nasal cannula (Fisher & Paykel healthcare, New Zealand) with flow 10l/min
Other: 30l/min — For inhalation was used diethilene penta-acetic triamine technetium (99mTc-DTPA) with radioactivity of 1 millicuries (Noble et al., 2007) and 0.9% saline solution with a total volume of 1 ml using vibrating mesh inhaler (Aerogen Ltd, Galway , Ireland) with the respiratory care system for the high flow ( Fisher & Paykel healthcare, New Zealand) and nasal cannula (Fisher & Paykel healthcare, New Zealand) with flow 30l/min.
Other: 50l/min — For inhalation was used diethilene penta-acetic triamine technetium (99mTc-DTPA) with radioactivity of 1 millicuries (Noble et al., 2007) and 0.9% saline solution with a total volume of 1 ml using vibrating mesh inhaler (Aerogen Ltd, Galway , Ireland) with the respiratory care system for the high flow ( Fisher & Paykel healthcare, New Zealand) and nasal cannula (Fisher & Paykel healthcare, New Zealand) with flow 50l/min.

SUMMARY:
The aerosol associated with noninvasive ventilation (NIV) and high flow therapy with nasal interface have been employed in an attempt to relieve respiratory distress and optimize the deposition of drugs by inhalation.

Some studies report the effects of NIV association with fogging in healthy subjects, asthmatics and COPD 7.8, but studies evaluating the association between high flow nasal mist interface and therapy are scarce and most are found in vitro and animal models. The objective of this study is to evaluate the deposition of the aerosol scintigraphy using the high flow nasal interface system with vibrating mesh nebulizers using in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* The study included healthy individuals of both sexes,
* between 18 to 65 years,
* without history of lung disease and forced vital capacity (FVC) or forced expiratory volume in the first second (FEV1) higher or equal to 80% from predicted values,
* ability to verbal commands understand and
* willing to provide signed consent to participate in this study.

Exclusion Criteria:

* Participants were excluded if there unable to understand and follow the procedures and were pregnant and unable to tolerate nebulization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
radioaerosol deposition index into the lungs | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Alcoforado, MsC, Principal Investigator — UFPE
Locations (1):
- Laboratório de Fisiologia e Fisioterapia Cardiopulmonar, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Alcoforado L, Ari A, Barcelar JM, Brandao SCS, Fink JB, de Andrade AD. Impact of Gas Flow and Humidity on Trans-Nasal Aerosol Deposition via Nasal Cannula in Adults: A Randomized Cross-Over Study. Pharmaceutics. 2019 Jul 7;11(7):320. doi: 10.3390/pharmaceutics11070320. PMID 31284680